CLINICAL TRIAL: NCT07113665
Title: Phase I Trial of MR-guided Focused Ultrasound (MRgFUS) Bilateral Capsulotomy for the Treatment of Refractory Anorexia Nervosa With Co-morbid Obsessive Compulsive Disorder or Major Depressive Disorder
Brief Title: Magnetic Resonance-Guided Focused Ultrasound Bilateral Capsulotomy for Refractory Anorexia Nervosa With Comorbid Obsessive Compulsive Disorder or Major Depressive Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6590
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa (DSM-IV Revised Criteria)
Keywords: Anorexia Nervosa; MR-guided Focused Ultrasound; bilateral capsulotomy; Obsessive Compulsive Disorder; Major Depressive Disorder
MeSH Terms: conditions — Anorexia Nervosa; Obsessive-Compulsive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR- guided Focused Ultrasound Capsulotomy (Experimental): Participants in this arm will undergo a single MRI-guided focused ultrasound (MRgFUS) thermal ablation procedure targeting the anterior limb of the internal capsule (ALIC). The procedure is performed using the ExAblate 4000 MRgFUS system, with real-time MR thermometry to ensure precise lesioning.
  This intervention is intended for individuals with treatment-refractory anorexia nervosa (AN) and comorbid obsessive-compulsive disorder (OCD) and/or major depressive disorder (MDD) who meet surgical eligibility criteria. All participants will complete standardized psychiatric and quality of life assessments at baseline and follow-up time points up to 24 months post-treatment to evaluate safety, feasibility, and preliminary clinical efficacy.
  Interventions: Device: ExAblate Neuro 4000

INTERVENTIONS:
Device: ExAblate Neuro 4000 — The ExAblate Neuro 4000 is an MRI-guided focused ultrasound (MRgFUS) system designed to perform noninvasive thermal ablation of targeted brain tissue. In this study, the ExAblate Neuro 4000 will be used to perform a bilateral capsulotomy by ablating the anterior limb of the internal capsule (ALIC) in patients with treatment-refractory anorexia nervosa (AN) and comorbid obsessive-compulsive disorder (OCD) and/or major depressive disorder (MDD). The procedure will be conducted under real-time MRI guidance and thermometry to ensure accurate targeting and controlled thermal delivery. This study aims to evaluate the safety, feasibility, and preliminary clinical benefit of MRgFUS in improving psychiatric symptoms and quality of life in this patient population.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and initial clinical effectiveness of MRI-guided focused ultrasound (MRgFUS) thermal ablation (capsulotomy) in patients with treatment-refractory anorexia nervosa (AN) and comorbid obsessive-compulsive disorder (OCD) and major depressive disorder (MDD). The main questions it aims to answer are:

1. Can MR-guided focused ultrasound capsulotomy be safely delivered through an intact skull in patients with treatment-refractory anorexia nervosa and comorbid OCD and/or MDD, with a safety and side-effect profile comparable to traditional radiofrequency neurosurgical approaches?
2. Does MRgFUS capsulotomy produce clinical outcomes comparable to open surgical ablative procedures-specifically, improvements in anxiety, mood, quality of life, anorexia nervosa psychopathology, habit formation, and weight-in patients with treatment-refractory anorexia nervosa?

Participants will:

1. Undergo baseline imaging and clinical assessments
2. Receive a single MRgFUS capsulotomy targeting the ALIC
3. Be monitored for 24 months post-treatment to assess adverse events, quality of life, and symptom changes using standardized clinical and neuropsychiatric measures

DETAILED DESCRIPTION:
This is a single-centre, prospective, single-arm, non-randomized Phase I study evaluating the safety, feasibility, and preliminary clinical benefit of MRI-guided focused ultrasound (MRgFUS) for the treatment of treatment-refractory anorexia nervosa (AN) with comorbid obsessive-compulsive disorder (OCD) and/or major depressive disorder (MDD).

A total of 10 patients will be enrolled and treated with a single MRgFUS capsulotomy targeting the anterior limb of the internal capsule (ALIC).

Participants will undergo comprehensive pre-treatment evaluations, including psychiatric assessment, physical and nutritional status review, MRI imaging, and surgical eligibility screening. The treatment will be performed using the ExAblate 4000 system under continuous MRI guidance and real-time thermometry.

Participants will be followed at regular intervals, including immediately post-treatment and at 1, 3, 6, 12, 18, and 24 months post-procedure, to evaluate safety and changes in clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 and ≤65 years of age, inclusive.
2. Patients who are competent and willing to give consent and able to attend study visits, as determined by both study Psychiatrist and the surgeon.
3. DSM-V diagnosis of Anorexia Nervosa, with co-morbid diagnosis of OCD and/or Major depressive disorder.
4. Treatment refractoriness indicated by any of:

   1. Duration of illness more than 10 years with no more than three months of remission in terms of weight;
   2. At least three attempts at expert hospital based treatment that were not successful or where there was no sustained response to treatment;
   3. A pattern of increased medical instability requiring at least two episodes of emergency/involuntary re-feeding and lasting at least two years;
5. Ability to provide informed consent/competent to make medical decisions.

Exclusion Criteria:

1. Patients with unstable cardiac status [e.g. Unstable angina pectoris on medication, Patients with documented myocardial infarction within six months, Congestive heart failure requiring medication (other than diuretic), Patients on anti-arrhythmic drugs, Severe hypertension (diastolic BP > 100 on medication)]
2. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
3. Laboratory biochemical evidence of abnormal bleeding and/or coagulopathy, including risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter or abnormal INR)
4. Cerebrovascular disease (e.g. CVA within 6 months) or history of intracranial hemorrhage
5. Untreated, uncontrolled sleep apnea
6. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
7. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment
8. Are participating or have participated in another clinical trial in the last 30 days
9. Patients unable to communicate with the investigator and staff.
10. Presence of significant cognitive impairment
11. History of psychosis on clinical evaluation.
12. Patients with brain tumors already known or revealed on pretreatment MRI
13. Currently pregnant (as determined by history and serum HCG) or lactating.
14. Chemical abuse or dependence within the previous six months
15. Presence of a metabolic pathology interfering with eating or digestion (e.g. diabetes).
16. Body mass index (BMI) less than 13

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Safety and Feasibility of MRgFUS Capsulotomy in Patients with Treatment-Refractory Anorexia Nervosa | From day of treatment through 24 months post-treatment with evaluations at immediate post-op, 1, 3, 6, 12, 18 and 24 months.
  The frequency and severity of adverse events associated with ExAblate Transcranial Magnetic Resonance-guided Focused Ultrasound (MRgFUS) will be evaluated in patients with treatment-refractory anorexia nervosa and comorbid obsessive-compulsive disorder (OCD) and/or major depressive disorder (MDD). All adverse events-including procedure-related complications, neurological events, and other safety concerns-will be systematically documented, monitored, and assessed throughout the study duration.

SECONDARY OUTCOMES:
Change in Body Mass Index Following MRgFUS Capsulotomy | Assessments will be conducted at baseline, 1, 3, 6, 12, 18, and 24 months following the procedure.
  Body Mass Index (BMI) will be used as an objective indicator of weight change and nutritional status. BMI will be calculated using weight (kg) divided by height (m²). Participants' BMI will be tracked over time to evaluate whether MRgFUS targeting the anterior limb of the internal capsule (ALIC) is associated with weight stabilization or improvement in individuals with treatment-refractory anorexia nervosa.
  Recommended BMI (Body Mass Index) for most adults is generally:
  Underweight: Below 18.5 Normal/Healthy weight: 18.5 - 24.9 Overweight: 25.0 - 29.9 Obese: 30.0 and above
  Notes:
  1. The above mentioned ranges are from the World Health Organization (WHO) and are intended for adults 18-65 years old.
  2. BMI is a quick screening tool but doesn't account for muscle mass, bone density, age or gender.
Change in Depressive Symptoms Using the Beck Depression Inventory | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post-treatment.
  The Beck Depression Inventory (BDI) is a 21-item self-report inventory assessing the presence and severity of depressive symptoms. Each item is scored from 0 to 3, with a total score range of 0 to 63. Higher scores reflect more severe depressive symptoms.
Change in Anxiety Symptoms Using the Beck Anxiety Inventory | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post-treatment.
  Evaluate the effectiveness of MR-guided Focused Ultrasound (MRgFUS) in reducing anxiety symptom severity using the Beck Anxiety Inventory (BAI), a validated patient-reported scale. Assessments will occur at baseline and at specified follow-up visits. The BAI consists of 21 items measuring common symptoms of anxiety experienced over the past week. Each item is rated on a scale from 0 (not at all) to 3 (severely). Total scores range from 0 to 63, with higher scores indicating more severe anxiety symptoms
Change in Quality of Life Using the Quality of Life Enjoyment and Satisfaction Questionnaire | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post-treatment.
  The Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ-SF) is a 14-item self-report questionnaire evaluating life satisfaction across various domains (e.g., physical health, mood, work, social life). Items are scored from 1 (very poor) to 5 (very good) and converted to a percentage (0-100%).
Change in Obsessive-Compulsive Symptoms Using the Obsessive Compulsive Inventory | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post-treatment.
  Obsessive Compulsive Inventory (OCI) - The Obsessive Compulsive Inventory is a self-report questionnaire used to assess the severity of obsessive-compulsive symptoms across six domains: washing, checking, ordering, obsessing, hoarding, and mental neutralizing. It consists of items scored from 0 (not at all) to 4 (extremely), with total scores ranging from 0 (no symptoms) to 72 (most severe symptoms). Higher scores indicate a worse outcome (greater severity of obsessive-compulsive symptoms).
Change in Suicide Risk Using the Columbia-Suicide Severity Rating Scale | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post-treatment.
  Columbia-Suicide Severity Rating Scale (C-SSRS) - The Columbia-Suicide Severity Rating Scale is a clinician-administered tool that evaluates suicidal ideation and behavior, including the severity and intensity of thoughts and the presence of actual, interrupted, or aborted suicide attempts. Scores range from 0 (no suicidal ideation or behavior) to 25 (most severe), with higher scores indicating a worse outcome (greater suicidal risk).

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No